CLINICAL TRIAL: NCT05907876
Title: Karabuk University
Brief Title: Test-Retest Reliability Of UULEX In Patients With Stroke
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Fatma Hale Altınkaya, INVESTIGATOR, Karabuk University
Other Study IDs: KarabukUN
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Stroke
Keywords: STROKE; UULEX; UPPER EXTREMITY
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Functional Test — UULEX uses a table of horizontal parallel lines with 8 levels. Each level is 84 cm wide and 8 cm high. The distance between the levels is 15 cm. The subject is seated on a straight chair with his/her feet on the floor facing the wall with the UULEX table. He/she holds a bar weighing 0.2 kg and lifts the bar at hip level. Keeping his/her arms shoulder-width apart, he/she raises the bar to different levels of the chart. As a warm-up, he/she is instructed to raise the bar to the first level and hold this position for 2 minutes. Then the bar is moved to each level and the levels are increased for 1 minute. The starting and ending point of each level is the hip joint. As the exercise progresses each minute, the weight of the bar is increased by 0.5 kg up to a maximum of 2 kg. During the test, a subject can move up to a maximum of a 2kg bar in a maximum of 12 minutes. The subject is instructed to continue the test until limited by the occurrence of symptoms.

SUMMARY:
Hemiplegia refers to a complete paralysis involving one side of the arm, trunk and leg. Stroke causes loss of ability and leads to loss of functionality of daily life activities of individuals. Changes in the anatomy of the joint should be analysed for a better understanding of upper extremity problems, especially shoulder problems and pain after stroke. In recent years, the prevalence of shoulder pain in haemiplegic patients has ranged between 5% and 84%. Shoulder pain makes movements of the upper limb difficult and affects gait. Lack of active movement and spasticity is an important cause of shoulder pain. Pain and changes in muscle tone affect upper limb functionality by 30-66%. Improvement in shoulder pain with the recovery of upper extremity functions is important in returning the person to active life independently, as well as obtaining effective hand function. There are many clinical tests used to evaluate upper extremity functionality after haemiplegia. One of them, the Unassisted Upper Extremity Exercise Test (UULEX), is a performance test that evaluates upper extremity performance. The unsupported upper extremity exercise test (UULEX) is a simple, inexpensive field test developed to measure upper arm exercise capacity, but there are no reports on its reliability for use in patients with hemiplegia. The aim of our study was to determine the test-retest reliability of the UULEX in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Having had a stroke
* Diagnosis of haemiplegia after a previous stroke
* Being between 18-78 years old
* Volunteering to participate in the study

Exclusion Criteria:

* Presence of pain in the upper limbs or neck
* Cognitive disorders
* Presence of comorbidity affecting upper extremity and hand functions (carpal tunnel syndrome, trigger finger, impingement syndrome, thoracic outlet syndrome, lateral and medial epicondylitis)
* History of upper extremity surgery

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with stroke receiving rehabilitation services in a rehabilitation centre
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Upper Limb Functionality | First Day
  It will be evaluated using UULEX.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Hale Altınkaya, Study Chair — Karabuk University

IPD SHARING:
Plan to Share IPD: No